CLINICAL TRIAL: NCT00976521
Title: A 2x2 Factorial, Randomized, Multicenter, Single-Blind Evaluation of Intracoronary Abciximab Infusion and Aspiration Thrombectomy in Patients Undergoing Percutaneous Coronary Intervention for Anterior ST-Segment Elevation Myocardial Infarction
Brief Title: The INFUSE - Anterior Myocardial Infarction (AMI) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atrium Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 901
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2013-07-08 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-05

CONDITIONS: Acute Anterior Myocardial Infarction
MeSH Terms: conditions — Anterior Wall Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Local infusion, thrombus aspiration (Experimental): Local infusion of abciximab using the ClearWay™ RX Infusion Catheter following thrombus aspiration.
  Interventions: Drug: Abciximab local infusion; Procedure: Thrombus aspiration
- Local infusion, no aspiration (Experimental): Local infusion of abciximab using the ClearWay™ RX Infusion Catheter and no aspiration
  Interventions: Drug: Abciximab local infusion
- No local infusion, thrombus aspiration (Active Comparator): No local infusion of abciximab, thrombus aspiration.
  Interventions: Other: No local infusion; Procedure: Thrombus aspiration
- No local infusion, no aspiration (Active Comparator): No local infusion abciximab and no thrombus aspiration
  Interventions: Other: No local infusion

INTERVENTIONS:
Drug: Abciximab local infusion — Local infusion of abciximab using the ClearWay™ RX Infusion Catheter
  Arms: Local infusion, no aspiration; Local infusion, thrombus aspiration
Other: No local infusion — Intervention without local infusion
  Arms: No local infusion, no aspiration; No local infusion, thrombus aspiration
Procedure: Thrombus aspiration — Thrombus aspiration
  Arms: Local infusion, thrombus aspiration; No local infusion, thrombus aspiration

SUMMARY:
This is a multicenter, open-label, controlled, single-blind, randomized study with up to 452 subjects enrolled in up to 50 US and European sites. Subjects who present with anterior ST-elevation myocardial infarction (STEMI) and an occluded proximal or mid left anterior descending (LAD) with TIMI 0/1/2 flow will be eligible for randomization to one of the following arms:

1. Local infusion of abciximab following thrombus aspiration
2. Local infusion of abciximab and no thrombus aspiration
3. No local infusion and thrombus aspiration
4. No local infusion and no thrombus aspiration

In addition, a cardiac magnetic resonance imaging (MRI) sub-study evaluating microvascular obstruction (MVO) will be performed with up to 160 subjects at up to 20 sites.

DETAILED DESCRIPTION:
The primary objective of the study is to demonstrate that among subjects undergoing primary PCI for anterior STEMI treated with a bivalirudin monotherapy anticoagulation strategy, the intracoronary infusion of an abciximab bolus with or without thrombus aspiration prior to stent implantation, compared to no infusion with or without thrombus aspiration (standard of care), results in 1) reduced infarct size measured by cardiac MRI at 30 days (range -7 days/+14 days; i.e., between 23 and 44 days), 2) reduce microvascular obstruction (MVO) by cardiac MRI at 5 + 2 days (i.e., between 3 and 7 days), 3) enhanced ST-segment resolution, 4) improved myocardial perfusion, 5) reduced thrombus burden and angiographic complications, and 6) no increase in major and minor bleeding.

ELIGIBILITY:
Key Inclusion Criteria:

* The subject must be >18 years of age;
* Subject is experiencing clinical symptoms consistent with AMI (e.g., chest pain, arm pain, etc.,) >30 minutes duration and unresponsive to nitroglycerin;
* Anterior MI with ECG showing at least 1 mm of ST-segment elevation in 2 or more contiguous leads in V1-V4, or new (or presumably new) left bundle branch block;
* Anticipated symptom onset to balloon or aspiration time of ≤5 hours;
* The subject and his/her physician are willing to comply with specified follow-up evaluations;
* The subject or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided and signed written informed consent, approved by the appropriate Medical Ethics Committee (MEC) or Institutional Review Board (IRB)
* Infarct artery located in the proximal or mid left anterior descending coronary artery, with TIMI 0/1/2 flow at the time of initial diagnostic angiography (prior to wire passage);
* Based on coronary anatomy, PCI is indicated for revascularization;
* Only one epicardial coronary artery will be treated;
* Expected ability to deliver a ClearWay™ RX Infusion Catheter to the infarct lesion (absence of excessive tortuosity, diffuse disease or moderate/heavy calcification).

Key Exclusion Criteria:

* Prior myocardial infarction, or known prior systolic dysfunction (known ejection fraction <40% by any prior measure or regional wall motion abnormalities);
* An elective surgical procedure is planned that would necessitate interruption of anti-platelet agents during the first twelve months post enrollment;
* Subjects who previously underwent coronary stent implantation and in whom coronary angiography demonstrates stent thrombosis to be the cause of the AMI;
* Subject has previously undergone an angioplasty or stenting procedure in the left anterior descending artery;
* Definite planned use of aspiration, atherectomy, thrombectomy and/or distal protection catheters prior to PTCA or stent implantation (other than in subjects randomized to thrombus aspiration);
* Any contraindication to undergo MRI imaging.
* Multivessel intervention required during the index procedure (subjects may be enrolled if treatment of more than one lesion in the LAD or its branches is required, however) (planned staged procedures are permitted with strong recommendation to be performed after 30-day clinical and MRI endpoints are completed);
* Severe vessel tortuosity, diffuse disease or severe calcification is present which may impede successful delivery of the ClearWay™ RX Infusion Catheter or the Export® Aspiration Catheter;
* Features are present highly unfavorable for PCI;
* Target lesion is present within a bypass graft conduit;
* MI is due to thrombosis within or adjacent to a previously implanted stent;
* Left ventriculography demonstrates severe mitral regurgitation or a VSD;
* Unprotected left main stenosis >40% or that will require intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2009-09; Primary Completion 2012-02 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg W Stone, MD, Principal Investigator — Columbia University
Locations (38):
- United States (7):
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Carolinas Medical Center-SHVI, Charlotte, North Carolina
  - Moses Cone Vascular Center, Greensboro, North Carolina
  - Geisinger Medical Center, Danville, Pennsylvania
  - Harrisburg Hospital/ Pinnacle Health, Harrisburg, Pennsylvania
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
- Austria (5):
  - Landeskrankenhaus Bruck/Mur, Bruck/Mur, Austria
  - Landeskrankenhaus Graz West, Graz, Austria
  - Univ. Klinik für Innere Medizin III Innsbruck, Innsbruck, Austria
  - Univ. Klinik für Innere Medizin II, Vienna, Austria
  - Landeskrankenhaus Braunau/Simbach, Braunau am Inn
- Germany (6):
  - Universitätsmedizin Mannheim - I. Medizinische Klinik, Mannheim, Germany
  - Klinikum der Universität Regensburg, Regensburg, Germany
  - Charite- University Medicine Campus Benjamin Franklin, Berlin
  - Klinikum Villingen Kardiologie, Darmstadt
  - Facharzt fur Innere Medizin/Kardiologie, Ludwigshafen
  - Universtitätsklinikuim Ulm, Ulm
- Netherlands (3):
  - Ziekenhuis Rijnstate, Arnhem, NL
  - Catharina Hospital Eindhoven, Eindhoven
  - Isala Klinieken, Locatie de Weezenlanden, Zwolle
- Poland (8):
  - Polsko - Amerykańskie Kliniki Serca II Oddział Kardiologiczny American Heart of Poland Sp. z o.o., Bielsko-Biala, Poland
  - Krakowski Szpital Specjalistyczny im. Jana Pawła II w Krakowie, Centrum Interwencyjne Leczenia Chorób Serca i Naczyń, Krakow, Poland
  - SPZOZ Szpital Uniwersytecki w Krakowie, Samodzielna Pracownia Hemodynamiki i Angiografii, Krakow, Poland
  - Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie Pracownia Hemodynamiki I Katedry i Kliniki Kardiologii, Warsaw, Poland
  - Instytut Kardiologii im. Prymasa Tysiąclecia Kardynała Stefana Wyszyńskiego,I Samodzielna Pracownia Hemodynamiki, Warsaw, Poland
  - Krakowskie Centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii, Krakow
  - Pracownia Hemodynamiki Oddziału Kardiologicznego Wojewódzkiego Centrum Medycyny w Opolu, Opole
  - Centrum Kardiologii Inwazyjnej GVM Carint, Oświęcim
- United Kingdom (9):
  - University Hospitals of Leicester - Glenfield Hospital, Leicester, U.k.
  - King's College Hospital, London, U.k.
  - Manchester Royal Infirmary, Manchester, U.k.
  - Wythenshawe Hospital, Manchester, U.k.
  - Southampton University Hospital, Southampton, U.k.
  - Royal Victoria Hospital, Belfast Trust, Belfast
  - Bristol Heart Institute, Bristol
  - Golden Jubilee National Hospital, Glasgow
  - Freeman Hospital, Newcastle upon Tyne

REFERENCES:
- [Derived] Giustino G, Redfors B, Brener SJ, Kirtane AJ, Genereux P, Maehara A, Dudek D, Neunteufl T, Metzger DC, Crowley A, Mehran R, Gibson CM, Stone GW. Correlates and prognostic impact of new-onset heart failure after ST-segment elevation myocardial infarction treated with primary percutaneous coronary intervention: insights from the INFUSE-AMI trial. Eur Heart J Acute Cardiovasc Care. 2018 Jun;7(4):339-347. doi: 10.1177/2048872617719649. Epub 2017 Aug 22. PMID 28828881
- [Derived] Tomey MI, Mehran R, Brener SJ, Maehara A, Witzenbichler B, Dizon JM, El-Omar M, Xu K, Gibson CM, Stone GW. Sex, adverse cardiac events, and infarct size in anterior myocardial infarction: an analysis of intracoronary abciximab and aspiration thrombectomy in patients with large anterior myocardial infarction (INFUSE-AMI). Am Heart J. 2015 Jan;169(1):86-93. doi: 10.1016/j.ahj.2014.06.019. Epub 2014 Jul 3. PMID 25497252
- [Derived] Guerchicoff A, Brener SJ, Maehara A, Witzenbichler B, Fahy M, Xu K, Gersh BJ, Mehran R, Gibson CM, Stone GW. Impact of delay to reperfusion on reperfusion success, infarct size, and clinical outcomes in patients with ST-segment elevation myocardial infarction: the INFUSE-AMI Trial (INFUSE-Anterior Myocardial Infarction). JACC Cardiovasc Interv. 2014 Jul;7(7):733-40. doi: 10.1016/j.jcin.2014.01.166. PMID 25060015
- [Derived] Stone GW, Witzenbichler B, Godlewski J, Dambrink JH, Ochala A, Chowdhary S, El-Omar M, Neunteufl T, Metzger DC, Dizon JM, Wolff SD, Brener SJ, Mehran R, Maehara A, Gibson CM. Intralesional abciximab and thrombus aspiration in patients with large anterior myocardial infarction: one-year results from the INFUSE-AMI trial. Circ Cardiovasc Interv. 2013 Oct 1;6(5):527-34. doi: 10.1161/CIRCINTERVENTIONS.113.000644. Epub 2013 Oct 1. PMID 24084626
- [Derived] Brener SJ, Maehara A, Dizon JM, Fahy M, Witzenbichler B, Parise H, El-Omar M, Dambrink JH, Mehran R, Oldroyd K, Gibson CM, Stone GW. Relationship between myocardial reperfusion, infarct size, and mortality: the INFUSE-AMI (Intracoronary Abciximab and Aspiration Thrombectomy in Patients With Large Anterior Myocardial Infarction) trial. JACC Cardiovasc Interv. 2013 Jul;6(7):718-24. doi: 10.1016/j.jcin.2013.03.013. PMID 23866184
- [Derived] Brener SJ, Witzenbichler B, Maehara A, Dizon J, Fahy M, El-Omar M, Dambrink JH, Genereux P, Mehran R, Oldroyd K, Parise H, Gibson CM, Stone GW. Infarct size and mortality in patients with proximal versus mid left anterior descending artery occlusion: the Intracoronary Abciximab and Aspiration Thrombectomy in Patients With Large Anterior Myocardial Infarction (INFUSE-AMI) trial. Am Heart J. 2013 Jul;166(1):64-70. doi: 10.1016/j.ahj.2013.03.029. Epub 2013 Apr 30. PMID 23816023
- [Derived] Stone GW, Maehara A, Witzenbichler B, Godlewski J, Parise H, Dambrink JH, Ochala A, Carlton TW, Cristea E, Wolff SD, Brener SJ, Chowdhary S, El-Omar M, Neunteufl T, Metzger DC, Karwoski T, Dizon JM, Mehran R, Gibson CM; INFUSE-AMI Investigators. Intracoronary abciximab and aspiration thrombectomy in patients with large anterior myocardial infarction: the INFUSE-AMI randomized trial. JAMA. 2012 May 2;307(17):1817-26. doi: 10.1001/jama.2012.421. Epub 2012 Mar 25. PMID 22447888
- [Derived] Gibson CM, Maehara A, Lansky AJ, Wohrle J, Stuckey T, Dave R, Cox D, Grines C, Dudek D, Steg G, Parise H, Wolff SD, Cristea E, Stone GW. Rationale and design of the INFUSE-AMI study: A 2 x 2 factorial, randomized, multicenter, single-blind evaluation of intracoronary abciximab infusion and aspiration thrombectomy in patients undergoing percutaneous coronary intervention for anterior ST-segment elevation myocardial infarction. Am Heart J. 2011 Mar;161(3):478-486.e7. doi: 10.1016/j.ahj.2010.10.006. Epub 2011 Jan 28. PMID 21392601

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 28-Nov-09 and 02-Dec-11, 452 subjects meeting all clinical eligibility criteria were consented and enrolled at 37 US and European sites.
Pre-assignment Details: Subjects were randomized in a 1:1:1:1 ratio to each of the randomized groups (abciximab infusion with aspiration, abciximab infusion without aspiration, no infusion with aspiration, no infusion without aspiration).
Groups:
- Local Infusion, Thrombus Aspiration: Local infusion of abciximab using the ClearWay™ RX Infusion Catheter following thrombus aspiration.
  A 6 French Export® Aspiration Catheter is passed across the target coronary segment during continuous aspiration. Several passes should be made across the lesion to attempt to remove residual thrombus, always with continuous aspiration when advancing or withdrawing the catheter until the operator appreciates that no further thrombus is being removed.
  After withdrawing the aspiration catheter, the lesion is crossed with a 1.0 mm, 1.5 mm, or 2.0 mm diameter ClearWay™ RX Infusion Catheter (depending on the lumen diameter created by thrombus aspiration and the reference vessel diameter). If the lesion is successfully crossed or penetrated by at least 1 mm, an intracoronary bolus of abciximab (0.25 mg/kg body weight, given as 10 cc over approximately 60 seconds) is infused through the ClearWay™ RX Infusion Catheter.
- Local Infusion, no Aspiration: Local infusion of abciximab using the ClearWay™ RX Infusion Catheter and no thrombus aspiration.
  The initial device used to cross the lesion is a 1.0 mm or 1.5 mm diameter ClearWay™ RX Infusion Catheter (1.0 mm for complete occlusion).
  If the lesion is successfully crossed or penetrated by at least 1 mm, an intracoronary bolus of abciximab (0.25 mg/kg body weight, infused at a rate of 10 cc over approximately 60 seconds) is infused through the ClearWay™ RX Infusion Catheter.
- No Local Infusion, Thrombus Aspiration: No local infusion of abciximab, thrombus aspiration.
  A 6 French Export® Aspiration Catheter is passed across the target coronary segment during continuous aspiration. Several passes should be made across the lesion to attempt to remove residual thrombus, always with continuous aspiration when advancing or withdrawing the catheter until the operator appreciates that no further thrombus is being removed.
- No Local Infusion, no Aspiration: No local infusion of abciximab and no thrombus aspiration.
  The lesion is pre-dilated with at least a 2.0 mm angioplasty balloon and then stent implantation is performed as per standard of care.
Period: Overall Study
Arm/Group | Local Infusion, Thrombus Aspiration | Local Infusion, no Aspiration | No Local Infusion, Thrombus Aspiration | No Local Infusion, no Aspiration
Started | 118 | 111 | 111 | 112
Completed | 109 | 99 | 102 | 93
Not Completed | 9 | 12 | 9 | 19

BASELINE CHARACTERISTICS:
Groups:
- Local Infusion, no Aspiration: Local infusion of abciximab using the ClearWay™ RX Infusion Catheter and no thrombus aspiration
- No Local Infusion, no Aspiration: No local infusion of abciximab and no thrombus aspiration
- Total: Total of all reporting groups
Arm/Group | Local Infusion, Thrombus Aspiration | Local Infusion, no Aspiration | No Local Infusion, Thrombus Aspiration | No Local Infusion, no Aspiration | Total
Number analyzed (Participants) | 118 | 111 | 111 | 112 | 452
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 80 | 79 | 61 | 67 | 287
  >=65 years | 38 | 32 | 50 | 45 | 165
Age Continuous [Median (Inter-Quartile Range); unit: years] | 60.0 [52.0 to 66.0] | 56.0 [49.0 to 68.0] | 62.0 [53.0 to 73.0] | 62.5 [52.5 to 71.0] | 61.0 [52.0 to 72.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 27 | 26 | 31 | 118
  Male | 84 | 84 | 85 | 81 | 334
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 12 | 12 | 53
  Poland | 25 | 24 | 27 | 23 | 99
  Austria | 13 | 14 | 11 | 9 | 47
  Netherlands | 14 | 11 | 10 | 15 | 50
  Germany | 22 | 21 | 19 | 19 | 81
  United Kingdom | 30 | 26 | 32 | 34 | 122

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint - Infarct Size at 30 Days as a Percentage of Total Left Ventricular Mass - Abciximab Infusion vs. No Infusion
Description: The primary endpoint of the INFUSE AMI study is infarct size as a percentage of total left ventricular mass at 30 days as measured by cardiac MRI (cMRI), comparing the pooled randomized active (abciximab) infusion to the pooled non infusion arms, without regard to aspiration.
Time Frame: 30 Days Post Index Procedure
Population: Evaluable cardiac MRI (cMRI) results at 30 days to assess percentage of total left ventricular mass were available for 181 and 172 patients randomized to intracoronary abciximab infusion versus no abciximab infusion, respectively for the ITT (intention to treat) analysis set.
Measure: Median (Inter-Quartile Range); unit: Percentage of Left Ventricular Mass
Groups:
- Abciximab Infusion: Abciximab Infusion includes subjects randomized to either the following two arms: abciximab active infusion arm with aspiration or abciximab infusion arm without aspiration. If the lesion is successfully crossed or penetrated by at least 1 mm, an intracoronary bolus of abciximab (0.25 mg/kg body weight, given as 10 cc over approximately 60 seconds) is infused through the ClearWay™ RX Infusion Catheter.
- No Infusion: No Infusion includes subjects randomized to either the following two arms: no abciximab infusion with aspiration or no abciximab infusion without aspiration. If randomized to abciximab infusion with aspiration, a 6 French Export® Aspiration Catheter is passed across the target coronary segment during continuous aspiration. Several passes should be made across the lesion to attempt to remove residual thrombus, always with continuous aspiration when advancing or withdrawing the catheter until no further thrombus is being removed. If randomized to no abciximab infusion without aspiration, the lesion is pre-dilated with at least a 2.0 mm angioplasty balloon and then stent implantation is performed as per standard of care.
- Combined: Combined includes subjects randomized to all four arms.
Arm/Group | Abciximab Infusion | No Infusion | Combined
Number analyzed (Participants) | 181 | 172 | 353
Percentage of Left Ventricular Mass | 15.1 [6.8 to 22.7] | 17.9 [10.3 to 25.4] | 17.2 [7.4 to 23.6]
Statistical Analysis 1: Comparison: Abciximab Infusion vs No Infusion; The primary endpoint of infarct size at 30 days measured by cardiac MRI, was summarized using the median, IQR, minimum and maximum values, in each infusion group, comparing the pooled active infusion arm to the pooled control non-infusion arm with the Wilcoxon rank sum test in the ITT analysis set. Data was only analyzed in subjects completing the cardiac MRI study and for whom the imaging data was received and deemed analyzable by the core laboratory; Test type: Superiority or Other; p = 0.034, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Major Secondary Endpoint - Infarct Size at 30 Days as a Percentage of Total Left Ventricular Mass - Aspiration vs. No Aspiration
Description: The major secondary endpoint of the INFUSE AMI Study is infarct size as a percentage of total myocardial mass at 30 days measured by cardiac MRI (cMRI), comparing the pooled randomized aspiration arms to the pooled no aspiration arms, without regard to abciximab infusion.
Time Frame: 30 Days
Population: Evaluable cardiac MRI (cMRI) results at 30 days to assess percentage of total myocardial mass were available for 192 and 190 patients randomized to thrombus aspiration versus no no thrombus aspiration, respectively for the ITT (intention to treat) analysis set.
Measure: Median (Inter-Quartile Range); unit: Percentage of Total Myocardial Mass
Groups:
- Thrombus Aspiration: Thrombus aspiration includes subjects randomized to either the following two arms: abciximab active infusion arm with aspiration or no abciximab infusion with aspiration. A 6 French Export® Aspiration Catheter is passed across the target coronary segment during continuous aspiration. Several passes should be made across the lesion to attempt to remove residual thrombus, always with continuous aspiration when advancing or withdrawing the catheter. Multiple passes should be made with contrast injection after each pass until the operator appreciates that no further thrombus is being removed.
- No Aspiration: No aspiration includes subjects randomized to either the following two arms: abciximab infusion arm without aspiration or no abciximab infusion without aspiration. If randomized to abciximab infusion without aspiration, the lesion is successfully crossed or penetrated by at least 1 mm, an intracoronary bolus of abciximab (0.25 mg/kg body weight, infused at a rate of 10 cc over approximately 60 seconds) is infused through the ClearWay™ RX Infusion Catheter. If randomized to no abciximab without aspiration, the lesion is pre-dilated with at least a 2.0 mm angioplasty balloon and then stent implantation is performed as per standard of care.
Arm/Group | Thrombus Aspiration | No Aspiration | Combined
Number analyzed (Participants) | 192 | 190 | 382
Percentage of Total Myocardial Mass | 17.0 [9.0 to 22.8] | 17.3 [7.1 to 25.5] | 17.2 [7.4 to 23.6]
Statistical Analysis 1: Comparison: Thrombus Aspiration vs No Aspiration; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.51, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Local Infusion, Thrombus Aspiration | Local Infusion, No Aspiration | No Local Infusion, Thrombus Aspiration | No Local Infusion, No Aspiration
Serious Adverse Events (participants affected / at risk) | 31/118 | 31/111 | 35/111 | 41/112
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Local Infusion, Thrombus Aspiration (N=118) | Local Infusion, No Aspiration (N=111) | No Local Infusion, Thrombus Aspiration (N=111) | No Local Infusion, No Aspiration (N=112)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 7 (7) | 7 (8) | 6 (8) | 5 (6)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac aneurysm (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cardiac pseudoaneurysm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Congestive heart failure (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Coronary artery perforation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart block (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Heart failure (Cardiac disorders) | 2 (2) | 4 (4) | 4 (4) | 11 (15)
Interventricular septum rupture (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 2 (2) | 3 (3) | 3 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular arrhythmia NOS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Defect interventricular septum (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GI bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Retroperitoneal bleed (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Accidental death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac death (General disorders) | 5 (5) | 2 (2) | 2 (2) | 2 (2)
Chest pain (General disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Chest pain (non-cardiac) (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thoracic pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulcer (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection systemic (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Localized infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (2)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic stent-graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral intake reduced (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Somatoform disorder cardiovascular (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney dysfunction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood transfusion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Chemotherapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Coronary angioplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Implantable cardioverter defibrillator insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Percutaneous coronary intervention (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal dialysis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Resuscitation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sternotomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterial rupture (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Peripheral ischemia (Vascular disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any proposed manuscript or publication will be submitted to Sponsor and Lead PI for comment at least 60 days prior to release of that manuscript or publication. There will be no publicizing of any data or results without the Sponsor's prior written permission. The publishing party will make every reasonable attempt to incorporate comments received from the Sponsor during such 60-day period.